CLINICAL TRIAL: NCT03496272
Title: Atrial Fibrillation (AF) Cycle Length Measured on Transesophageal Echocardiography : a Feasible Parameter for Predicting the Recurrence of AF in Patients With AF Converted to Sinus Rhythm After DC Cardioversion
Brief Title: Atrial Fibrillation Cycle Length Measured on Transesophageal Echocardiography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Yong Hyun Park, Associate Professor, Pusan National University Yangsan Hospital
Other Study IDs: PNUYH-IRB-05-2016-154
Record Dates: First submitted 2018-04-05; First posted 2018-04-12 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: The atrial fibrillation cycle length (AFCL) measured by electrophysiologic study is well known parameter for the maintenance of sinus rhythm after DC cardioversion (DCCV) or ablation therapy. The aim of this study was to test whether a AFCL measured by transesophageal echocardiography (AFCLTEE) could predict the outcome after DCCV.

Methods: In 100 consecutive patients with non-valvular AF, TEE will be performed within 6 hours before DCCV. The AFCLTEE was measured by averaging 10 sequential peak to peak intervals of atrial fibrillary waves seen in the pulsed wave Doppler image on the left atrial appendage. The primary endpoint was AF free survival rate at 6 months after DCCV.

ELIGIBILITY:
Inclusion Criteria:

* atrial fibrillation

Exclusion Criteria:

* moderate or severe mitral stenosis
* prosthetic heart valve

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with non-valvular atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
AF free survival rate at 6 months after DCCV | 6 month
  Atrial fibrillation free state at 6 months after direct current cardioversion

CONTACTS AND LOCATIONS:
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, South Korea